CLINICAL TRIAL: NCT02333968
Title: Effects of a Multifaceted Teleguided Pain Care Program in Patients With Cancer Pain
Brief Title: Self-management Support in Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Atrium Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UM 2011-5079
Record Dates: First submitted 2014-12-29; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Pain
Keywords: Cancer pain; Self-management; Randomized controlled trial
MeSH Terms: conditions — Pain; Cancer Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Self-management support
  Interventions: Behavioral: Self-management support
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Self-management support — The 12-week intervention consists of an iPad application for patients that is connected to a web application for nurses. Every morning and evening patients register pain and related symptoms by use of a pain diary. Patients are also requested to register medication intake. Graphical feedback is provided based on registered pain scores and medication intakes. Patients receive education on causes and treatment of pain, symptoms that require action, and methods to better control pain. Patients communicate with nurses via text message functionality within the application. Specialized nurses remotely monitor and analyze the patients' situation once every workday. Nurses have the opportunity to collaborate with the treating physician, pain specialist or multidisciplinary team.
  Arms: Intervention group

SUMMARY:
Pain is a prevalent and distressing symptom in patients with cancer, having an enormous impact on functioning and quality of life. Integration of patient self-management and professional care by means of care technology provides new opportunities in the outpatient setting. In this project a technology based and nurse delivered multicomponent self-management support intervention has been developed. Important components include monitoring, feedback, education, and nurse support. Following feasibility evaluation, the primary aim of this randomized controlled trial is to assess the effect of the intervention regarding pain intensity and quality of life as compared to care as usual. Secondary outcomes of the effect evaluation are self-efficacy, knowledge, anxiety and depression, and pain medication use. Besides, a cost-evaluation and summative process evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Patients who are under (palliative) anti-tumour treatment in a day clinic or outpatient clinic, or patients who have no treatment options available anymore
* Cancer (treatment related) pain > 2 weeks
* Pain is defined as a patient reported pain score of 4 or more on a numerical rating scale (scale 0-10)
* Living at home

Exclusion Criteria:

* Expected life expectancy < 3 months
* Chronic non-cancer pain
* Known cognitive impairments
* Participation in other studies that interfere with this study
* Not being able to read and understand the Dutch language
* Reduced vision
* Non-reachable by phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity (Brief Pain Inventory - Short Form (BPI-SF) | 12 weeks
  As measured with the Brief Pain Inventory - Short Form (BPI-SF)
Change in cancer related quality of life (European Organisation for Research and Treatment of Cancer Quality of life Questionnaire (EORTC QLQ-C30 version 3) | 12 weeks
  As measured with the European Organisation for Research and Treatment of Cancer Quality of life Questionnaire (EORTC QLQ-C30 version 3)

SECONDARY OUTCOMES:
Change in self-efficacy (Chronic Pain Self-efficacy Scale (CPSS) | 12 weeks
  As measured with the Chronic Pain Self-efficacy Scale (CPSS)
Change in knowledge about cancer pain (Pain Knowledge Questionnaire (PKQ) | 12 weeks
  As measured with the Pain Knowledge Questionnaire (PKQ)
Change in anxiety and depression (Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  As measured with the Hospital Anxiety and Depression Scale (HADS)
Change in pain medication use (Brief Pain Inventory - Short Form (BPI-SF), a cost diary and a pharmacist's overview) | 12 weeks
  As measured with the Brief Pain Inventory - Short Form (BPI-SF), a cost diary and a pharmacist's overview

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Atrium Medical Center, Heerlen
  - Maastricht University Medical Center, Maastricht

REFERENCES:
- [Derived] Hochstenbach LM, Courtens AM, Zwakhalen SM, van Kleef M, de Witte LP. Self-management support intervention to control cancer pain in the outpatient setting: a randomized controlled trial study protocol. BMC Cancer. 2015 May 19;15:416. doi: 10.1186/s12885-015-1428-1. PMID 25986294